CLINICAL TRIAL: NCT02132052
Title: Defining Cognitive and Motor Phenotypes of Parkinson's Disease (PD) With Magnetoencephalography
Brief Title: Defining Phenotypes of Movement Disorders :Parkinson's Plus Disorders (PD), Essential Tremor (ET), Cortical Basal Degeneration (CBD), Multiple Systems Atrophy (MSA), Magnetoencephalography.
Acronym: PHENO
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0952
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Essential Tremor; Multiple System Atrophy; Corticobasal Degeneration; Supranuclear Palsy, Progressive; Parkinson Disease
Keywords: Essential Tremor; Multiple System Atrophy; Corticobasal Degeneration; Supranuclear Palsy, Progressive; Parkinson's Disease; PD
MeSH Terms: conditions — Essential Tremor; Multiple System Atrophy; Corticobasal Degeneration; Supranuclear Palsy, Progressive; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigators hypothesize that there are specific characteristic of each cognitive and motor condition that can be defined using brains scans.

DETAILED DESCRIPTION:
Specific Aim 1: Determine which features of resting Magnetoencephalography (MEG) brain activity most sensitively discriminate between PD with normal cognition, PD with mild cognitive impairment (MCI), and PD dementia (PDD). Investigators predict that frontal network slowing and connectivity will discriminate between normal cognition and MCI while visuospatial network involvement will distinguish the PDD group.

Specific Aim 2: Determine which features of resting MEG brain activity most sensitively discriminate PDD from Alzheimer's Disease. Investigators predict that PDD will be distinguished from Alzheimer's (AD) on the basis of increased network connectivity, particularly in frontal and visuospatial networks.

Specific Aim 3 Investigate how resting state MEG activity correlates with task related brain activity. Investigators predict that resting state slowing will be associated with decreased task related brain activity.

Specific Aim 4: Determine which features of resting MEG brain activity most sensitively discriminate between motor subtypes of PD and also other relevant clinical populations (essential tremor and Parkinson plus syndromes). Investigators predict that frontal and parietal slowing and connectivity will discriminate PD from related conditions and that patterns of motor cortex connectivity and activity will differentiate among PD motor phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be age 40 or older,
* Be on stable medications for at least 30 days
* Montreal Cognitive Assessment (MOCA) of 26 or higher
* Scores within 1.5 standard deviations of age-matched norms for all neuropsychological tests
* Parkinson's Plus Disorders (PD) will be defined using United Kingdom (UK) Brain Bank Criteria.
* PD dementia (PDD) will be defined using the Movement Disorder Task Force 2007 criteria and supported by scores less than 1.5 standard deviations of age-matched norms in at least two domains.
* Probable Alzheimer's Disease (AD) will be defined using the National Institute on Aging-Alzheimer Association 2011 guidelines.
* Parkinson's Plus Disorders (PD) with mild cognitive impairment (MCI) will be defined by history, MOCA of 21 or higher, at least one score less than 1.5 standard deviations of age-matched norms, and cannot meet diagnostic criteria for PDD.
* Essential tremor and Parkinson plus syndromes (multiple systems atrophy, corticobasal degeneration, progressive supranuclear palsy) will be defined using previously published research criteria.19-22

Exclusion Criteria

* Features suggestive of other causes of parkinsonism/Parkinson-plus syndromes;
* Features suggestive of other causes of dementia, including moderate to severe cerebrovascular disease by history, or imaging or history of major head trauma;
* History of deep brain stimulation, ablation surgery, or other brain surgery;
* Evidence for depression based on the Hospital Anxiety Depression Scale (score > 11).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Colorado Hospital Movement Disorders Clinic Patients
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Focal oscillatory activity | May 2014
  Focal oscillatory activity: Focal band power for delta (0.5-4Hz), theta (4-8 Hz), alpha (9- 13 Hz), low beta (13-20 Hz), high beta (20-30 Hz) and gamma (30-50 Hz) activity will be derived from the autoregressive models.

SECONDARY OUTCOMES:
Spectral coherence: | May 2014
  2) Spectral coherence: Coherence is a measure of interdependence between two time series and can be applied to MEG data to determine functional networks.4a-chen Coherence will be derived from the autoregressive models.
Spectral Granger analysis: | May 2014
  3) Spectral Granger analysis: Granger analysis is a measure of the directionality of the relationship of two time series and can be applied to sensors or sources found to have significant coherence.
Reactivity: | May 2014
  Reactivity: Reactivity refers to changes in oscillatory activity between the eye open and eye closed conditions. Prior research in AD has shown significantly reduced reactivity compared to age-matched controls.
Complex network analysis: | May 2014
  Complex network analysis: Complex network analysis, originally developed in graph theory, is an approach to the study of complex systems such as brain networks. It allows investigators to characterize brain networks with a small number of neurobiologically meaningful and easily computable measures, including transitivity, global efficiency, and betweenness. These measures will be used to reveal the hypothesized connectivity abnormalities in PD and to differentiate different cognitive phenotypes in PD.

CONTACTS AND LOCATIONS:
Overall Officials: benzi Kluger, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University Of Colorado. Denver, MEG Lab, Aurora, Colorado, United States